CLINICAL TRIAL: NCT07327593
Title: Exercise Induced Hypoalgesia in Pain-free Stroke and Healthy Populations: a Cohort Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Neuron, Spain (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NeuronRehab
Record Dates: First submitted 2025-12-26; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Stroke; Pain; Exercise Induced Hypoalgesia
Keywords: Stroke; Pain; Exercise induced hypoalgesia; Cardiovascular training
MeSH Terms: conditions — Stroke; Pain

STUDY DESIGN:
Intervention Model Description: Two groups will be created (healthy and post-stroke). Both will carry out the same evaluation and exercise protocol to study the differences between both cohorts
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Outcome assessors will be blinded to intervention. Care providers will be blinded to the evaluation data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy cohort (Active Comparator): Age > 18 years; no neurological damage; no medical conditions that could affect the test; no pain of duration > 1 week in the 3 months preceding the enrollment. No serious medical conditions.
  First, pressure pain thresholds and conditioned pain modulation will be assessed. Then, participants will conduct a cardiovascular training for 30 minutes, and will be reassessed inmediately post-training and 30 minutes after.
  Interventions: Other: Cardiovascular training
- Post-stroke pain free cohort (Experimental): Ischemic or hemorrhagic stroke (> 3 months); older than 18 years old; of duration > 1 week in the 3 months preceding the enrollment. No other serious medical conditions.
  Post-stroke participants will get the same study protocol than healthy cohort.
  Interventions: Other: Cardiovascular training

INTERVENTIONS:
Other: Cardiovascular training — The cardiovascular training protocol will consist of a 5-minute warm-up aimed at reaching 70% of maximum heart rate (MHR) followed by 20 minutes of sustained work at this intensity (since maintaining this intensity is difficult, especially in the stroke cohort, we will allow for a margin of ±2-3% of MHR and provide feedback to increase or decrease the heart rate). We will aim to keep the heart rate below 73% of maximum heart rate, maintain blood pressure within safe ranges, and keep the effort level between 14/20 and 16/20

SUMMARY:
Exercise has shown multiple beneficial effects in both healthy and post-stroke populations. One of these is the acute reduction in sensitivity to painful stimuli, called exercise-induced hypoalgesia (EIH). This phenomenon has been studied since 1979 and has shown improvements in pain thresholds with both aerobic and resistance training in healthy, pain-free populations and different chronic pain conditions.

Although there has been extensive research on EIH in healthy populations and those with chronic musculoskeletal pain, surprisingly little attention has been given to individuals with neurological pathologies. Chronic pain is found in more than 50% of patients after stroke, and 70% of affected individuals experience pain on daily activities. Reported prevalences of post-stroke pain (PSP) between different studies, but there is a general consensus that it is an underreported phenomenon. Patients with pain experience greater cognitive and functional decline, fatigue, depression and lower quality of life.

Multiple factors contribute to PSP, and various approaches exist to treat all the variables influencing it. This study aims to compare the effects of exercise on pain perception in healthy individuals and stroke patients without pain, using the same cardiovascular training protocol, to better understand the mechanisms of EIH and its maintenance after stroke, ultimately aiming to improve the treatment of people with stroke.

ELIGIBILITY:
Inclusion Criteria:

* Healthy cohort: Age > 18 years; no neurological damage; no medical conditions that could affect the test; no pain
* Post-stroke cohort: : Ischemic or hemorrhagic stroke (> 3 months); age > 18 years; no pain

Exclusion Criteria:

* Healthy cohort: Any medical condition that could affect the test; pain in any location, of duration > 1 week in the 3 months preceding the trial.
* Post-stroke cohort: Unable to participate in the test (no possibility of transfer or active pedaling); medical contraindication to cardiovascular training for any reason; inability to follow instructions or communicate sensations during training; other neurological pathology; cardiac pathology (unstable angina, arrhythmias, aortic or left ventricular problems, myocarditis, pericarditis); pulmonary pathology that affects the test (pulmonary embolisms, pulmonary hypertension, etc.); renal or metabolic problems (severe renal dysfunction, uncontrolled diabetes, etc.); acute infection or fever; neurosurgery within 6 weeks prior to inclusion in the study; pain in any location, lasting > 1 week in the 3 months prior to the trial.; use of beta-blockers, antidepressants, or any medication that may alter heart rate measurements

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Pressure pain thresholds | Before the cardiovacular training, inmediately after the training, and 30 minutes after
  Pressure pain thresholds (PPT) are the most used pain sensitivity measure for these paradigms, and represent a static measure of pain, indicating the basal state of pain perception. It is usually measured with an algometer, which is pressured into the body of the participant, who is informed to warn in the moment when pressure starts to be painful. EIH has shown little differences between local and general effects, so we will measure PPT in both rectus femoris (local effects) and first dorsal interosseous (general effects), marking the exact points for ensuring the replicability of the measure after the exercise program. In the post-stroke cohort, this assessment will be performed on the non-paretic side, so that the possible loss of sensitivity due to the condition does not influence the measurements.
Conditioned pain modulation | Before the cardiovascular training, inmediately after the training and 30 minutes after
  Conditioned pain comulation (CPM) is the terminology used to describe the effect of endogenous pathways to enhance or diminish the afferent noxious stimuli. For this assessment the "cuff test" methodology will be carried out over the healthy arm of post-stroke participants. This methodology employs a test stimulus (TS) using pressure pain threshold measurement. Subsequently, an inflatable pressure cuff is applied, and its pressure is increased until the patient reports a pain sensation of 6 out of 10. While the cuff is inflated, the pressure pain threshold measurement is repeated to obtain a a conditioned stimulus (CS). The test result is then calculated by subtracting the pressures obtained on the algometer, thus calculating the CS-TS difference.
  CPM will be measured in the dominant side in the healthy cohort and in the healthy side in the post-stroke cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Herrera Rojas, Physical Therapist, Principal Investigator — Neuron, Spain
Locations (1):
- Neuron Madrid Río, Madrid, Madrid, Spain